CLINICAL TRIAL: NCT06378203
Title: Rehabilitation in Muscular Dystrophies From the Hospital Facility to the Home: Pilot Project
Brief Title: Rehabilitation in Muscular Dystrophies From the Hospital Facility to the Home: Pilot Project [RIMUDI]
Acronym: RIMUDI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEDEA 1013
Record Dates: First submitted 2024-03-19; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Muscular Dystrophies; Limb Girdle Muscular Dystrophy; Facio-Scapulo-Humeral Dystrophy; Becker Muscular Dystrophy
Keywords: muscular dystrophy; muscular training; muscular exercise; tele monitoring; home rehabilitation
MeSH Terms: conditions — Muscular Dystrophies; Muscular Dystrophies, Limb-Girdle; Muscular Dystrophy, Facioscapulohumeral; Muscular Dystrophy, Duchenne

STUDY DESIGN:
Intervention Model Description: Each patient will carry out a series of evaluation and training sessions (15 sessions) with a physiotherapist for the drafting of a personalized treatment plan which will subsequently be carried out "independently" at domicile.
  The home therapeutic proposal will include the use of the tele-rehabilitation system with virtual reality Home Kit - Virtual Reality Rehabilitation System (VRRS KHYMEIA) which allows to perform personalized games at home
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Limb GIrdle Muscular Dystrophy (Experimental): Open label study one arm
  Interventions: Other: tele-rehabilitation system with virtual reality Home Kit - Virtual Reality Rehabilitation System (VRRS KHYMEIA)

INTERVENTIONS:
Other: tele-rehabilitation system with virtual reality Home Kit - Virtual Reality Rehabilitation System (VRRS KHYMEIA) — A personalized exercise plan following macro-areas of objectives:
  * maintenance of muscle lengths with selective and/or prolonged static stretching exercises;
  * maintenance/improvement of muscle trophism with selective and/or postural and/or functional muscle recruitment exercises at moderate intensity (approximately 65%-70% of the maximum);
  * maintenance of respiratory muscle weakness with thoracic and/or diaphragmatic breathing exercises combined with muscle exercise;
  * endurance training with walking, cycle ergometer (to be used with both the upper and lower limbs) and treadmill at moderate intensity (approximately 65%-70% of the maximum).
  Home treatment will mostly take place with the KHYMEIA tele-rehabilitation system.

SUMMARY:
Until twenty years ago physical exercise in muscular dystrophies was considered harmful to the muscle cells, inducing an acceleration of cell necrosis. In fact, it is now certain and validated that an active lifestyle and the practice of controlled and regular physical activity are to be considered therapeutic in neuromuscular pathologies with the aim of optimizing muscular and cardio-respiratory function and preventing atrophy In particular, it seems that the optimal care is extensive and can be carried out in a safe and controlled manner even at home.

It is well documented that exercise has beneficial effects on muscle with increased strength and muscular endurance.

DETAILED DESCRIPTION:
This project was born precisely from the idea of giving an answer to the needs of patients on the one hand regarding being educated to carry out a physical activity/exercise "suitable" for the dystrophic muscle fiber and on the other to be able to insert this into everyday life activities, with remote expert monitoring.

One aim is to offer continuity of care between the hospital structure and the home, also offering a concrete response to the inconsistent care guaranteed for these chronic developmental diseases by the National Health Service. The drafting of a personalized therapeutic plan, to be implemented within the home, would not only support the patient's motor needs, but would also guarantee a positive impact on a psychological level, strengthening the patient's participation in shared therapeutic objectives and awareness of the same. This pilot project aims to evaluate the effectiveness of a 6-month tele-rehabilitation program for continuity of care in a population of subjects suffering from neuromuscular pathology. The primary outcome will then be integrated with an assessment of tolerance of the path and usability and acceptability of the tele-rehabilitation system used.

Each patient will carry out a series of evaluation and training sessions (15 sessions) with a physiotherapist for the drafting of a personalized treatment plan that subsequently will be carried out "independently" at domicile.

During these days, periodic clinical-instrumental evaluations indicated by the specific guidelines for each form of dystrophy and in particular cardiorespiratory and nutritional status ones will also be carried out.

Furthermore, "educational" support will also take place, instructing the patient about the benefits of maintaining an active lifestyle and regular practice of controlled physical activity.

The home therapeutic proposal will include the use of the tele-rehabilitation system with virtual reality Home Kit - Virtual Reality Rehabilitation System (VRRS KHIMEYA) which allows to perform personalized games at home.

ELIGIBILITY:
Inclusion Criteria:- definite genetic diagnosis of Limb Girdle Muscular Dystrophy: LGMD2A/R1(calpain 3 deficiency), LGMD2B/R2(dysferlin deficiency), LGMD2I/R9 (FKRP), LGMD2L /R11(ANOCTAMIN 5) or Facio Scapulo Humeral Dystrophy (FSHD) or Becker muscular dystrophy (BMD);

* strength values at the level of the main antigravity muscles > or equal to 3, according to the Medical Research Council (MRC) scale;
* independent walking in a protected (internal) environment, even with assistance;
* patients must have performed at least 1 clinical-functional evaluation at our facility in the year preceding the start of the trial.
* They must express compliance with joining the project and must not be followed from a physiotherapeutic point of view elsewhere during the 6 months of participation in the project.

Exclusion Criteria:

* dilated or ischemic heart disease with Left Ventricle Ejection Fraction <50%;
* chronic respiratory failure with Forced Vital Capacity < 40% predicted, nocturnal oxygen desaturation - > 5% of nocturnal time spent with peripheral oxygen saturation levels < 90).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
6 minute walk test (6MWT) | 6 months : Modification from month 0 (baseline) to month 6
  6 Minute Walk Test (measured in meters- normal range 500-600 meters in 6 minutes)
Motor Function Measure scale (MFM) | 6 months: Modification from month 0 (baseline) to month 6
  MFM measures Motor function at 3 levels (D1 change position and transfers; D2 axial and proximal motor function; D3 distal motor function), Each i item is scored on a 4-point Likert scale from 0 (cannot initiate the task) to 3 (performs the task fully). Item scores are summed, and the raw score is transformed to an overall total score ranging from 0 (severe functional impairment) to 100 (no functional impairment). rated in % from 0 to 100 and an overall percentage is calculated , in %)
Performance of Upper Limb (PUL) | 6 Months: Modification from month 0 (baseline) to month 6
  Performance of upper limb is a scale specifically designed to measure upper limb function in muscular dystrophy; there is an entry level item ranging from 0 to 6; the PUL scale test the proximal to distal progression of muscle weakness through three levels: high (shoulder domain), mid (elbow domain), and distal (wrist and finger domain); the PUL score (version 1.2) includes 22 items ; the overall scores ranges from 0 to 42
Time up and go (TUG) | 6 months: Modification from month 0 (baseline) to month 6
  Recording of the time required to stand up from a chair, walk for 3 meters and going back to the sitting position- normal range < 10 seconds

SECONDARY OUTCOMES:
Modification of fatigue and quality of life scales from T0 to T6 | 6 months: Modification from month 0 (baseline) to month 6
  Modified Fatigue Impact Scale (MFIS) composed by 3 sub scales (physical scale score final range from 0 to 36; COGNITIVE final range from 0 to 40; PSYCHOSOCIAL, final range score from 0 to 8) and 1 final total score ranging from 0 to 84
Short Form 36 (SF36) | 6 months: Modification from month 0 (baseline) to month 6
  one multi-item scale that assesses eight health concepts: 1) limitations in physical activities because of health problems; 2) limitations in social activities because of physical or emotional problems; 3) limitations in usual role activities because of physical health problems; 4) bodily pain; 5) general mental health (psychological distress and well-being); 6) limitations in usual role activities because of emotional problems; 7) vitality (energy and fatigue); and 8) general health perceptions. Each item with a score ranging from 0 to 100

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific Institute IRCCS Eugenio Medea, Bosisio Parini, Lecco, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Preisler N, Orngreen MC. Exercise in muscle disorders: what is our current state? Curr Opin Neurol. 2018 Oct;31(5):610-617. doi: 10.1097/WCO.0000000000000597. PMID 30036194
- [Background] Veenhuizen Y, Cup EHC, Jonker MA, Voet NBM, van Keulen BJ, Maas DM, Heeren A, Groothuis JT, van Engelen BGM, Geurts ACH. Self-management program improves participation in patients with neuromuscular disease: A randomized controlled trial. Neurology. 2019 Oct 29;93(18):e1720-e1731. doi: 10.1212/WNL.0000000000008393. Epub 2019 Sep 30. PMID 31570565
- [Background] Siciliano G, Simoncini C, Giannotti S, Zampa V, Angelini C, Ricci G. Muscle exercise in limb girdle muscular dystrophies: pitfall and advantages. Acta Myol. 2015 May;34(1):3-8. PMID 26155063
- [Background] Eagle M. Report on the muscular dystrophy campaign workshop: exercise in neuromuscular diseases Newcastle, January 2002. Neuromuscul Disord. 2002 Dec;12(10):975-83. doi: 10.1016/s0960-8966(02)00136-0. No abstract available. PMID 12467755
- [Background] Heutinck L, Jansen M, van den Elzen Y, van der Pijl D, de Groot IJM. Virtual Reality Computer Gaming with Dynamic Arm Support in Boys with Duchenne Muscular Dystrophy. J Neuromuscul Dis. 2018;5(3):359-372. doi: 10.3233/JND-180307. PMID 29991140
- [Background] Jansen M, de Groot IJ, van Alfen N, Geurts ACh. Physical training in boys with Duchenne Muscular Dystrophy: the protocol of the No Use is Disuse study. BMC Pediatr. 2010 Aug 6;10:55. doi: 10.1186/1471-2431-10-55. PMID 20691042